CLINICAL TRIAL: NCT07046377
Title: Comparative Study Between Adductor Canal Block Combined With (IPACK) Block Versus Genicular Nerves Block Combined With (IPACK) Block Regarding Postoperative Analgesic Effect After Knee Replacement Surgery.
Brief Title: Comparison Between Two Blocks in Analgesia After Knee Arthroplasty
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: FMASU MS64/2025
Record Dates: First submitted 2025-05-06; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-05

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Active Comparator): Adductor canal block + IPACK group
  Interventions: Procedure: ACB - IPACK
- Group 2 (Active Comparator): Genicular nerves block + IPACK block.
  Interventions: Procedure: GNB - IPACK

INTERVENTIONS:
Procedure: ACB - IPACK — will receive spinal anesthesia and ultrasound-guided Adductor canal nerve block, as well as infiltration of the space between the popliteal artery and the capsule of the posterior knee (IPACK) block.
  Arms: Group 1
Procedure: GNB - IPACK — will recieve spinal anesthesia and US guided Genicular nerves block and IPACK block.
  Arms: Group 2

SUMMARY:
Comparative Study between Adductor canal block combined with infiltration OF The interspace between popliteal artery and the capsule of the knee block versus genicular nerves Block combined with IPACK in Postoperative analgesia after knee replacement surgery

DETAILED DESCRIPTION:
Patient informed written consent and ethical committee approval of Faculty of Medicine; Ain Shams University will be obtained before patient allocation.

• Study procedures: Supervisors and experts will do all the study procedures.

Patients undergoing unilateral Total knee replacement (TKR) will be randomly assigned into one of the following groups using computer generated codes (15 patients in each group):

Group 1 (ACB - IPACK group): will receive spinal anesthesia and ultrasound-guided Adductor canal nerve block, as well as infiltration of the space between the popliteal artery and the capsule of the posterior knee (IPACK) block.

Group 2 (GNB - IPACK group): will recieve spinal anesthesia and US guided Genicular nerves block and IPACK block.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-85 years.
* Both sexes.
* American Society of Anesthesiologists (ASA) Physical Status Class I to III.
* Patients scheduled for unilateral TKA under spinal anesthesia.

Exclusion Criteria:

* Patient's refusal.
* American Society of Anesthesiologists (ASA) Physical Status Class above III.
* local infection.
* History of allergy to the medications used in the study. 5. Psychiatric disorder.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-01-29 (Actual); Primary Completion 2025-07-29 (Estimated); Study Completion 2025-07-29 (Estimated)

PRIMARY OUTCOMES:
1- Comparing both groups regarding the time needed ( in hours) for the first call rescue analgesia post operatively. | 5 minutes after ending of operation
  Total knee replacement (TKR) is a well-known popular surgical procedure for knee diseases, including end-stage knee osteoarthritis that causes severe postoperative pain and prolonged immobility.
  Acute pain control can be provided with multimodal analgesia, including non-steroidal anti-inflammatory drugs (NSAIDs) and opioids. However, NSAIDs cause many side effects as peptic ulcer and gastritis, also opioids have gastrointestinal side effects as constipation, nausea and vomiting as well as respiratory depression.
  Regional analgesia has been used as another modality to provide sufficient perioperative pain relief with minimal opioid consumption to avoid it's adverse effects peripheral nerve blocks (PNBs) is a common practice in orthopedic surgery. PNBs provide excellent pain management after TKA, promote early mobilization, and reduce the consumption of opioids, the incidence of opioid-related adverse effects, and the hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Mai Ma Abd ElAziz, MBBCH, Principal Investigator — Ain Shams University; Mai Ma Abd ElAziz Ibrahim, MBBCH, Principal Investigator — Ain Shams University
Locations (1):
- Ain shams university, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All data will be shared once Study is completed
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Before 1/2026
Access Criteria: Free